CLINICAL TRIAL: NCT06676644
Title: A Comparative Study on the Immunogenicity and Safety of Adjuvanted Versus Non-Adjuvanted Influenza Vaccines in the Elderly
Brief Title: Estimate the Safety and Effectiveness of Adjuvanted Influenza Vaccine Among Asian Elderly People When Compared to Non-adjuvanted Vaccines
Acronym: influenza
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Clinical Trial Center, Clinical professor, National Taiwan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 202409030MIND
Record Dates: First submitted 2024-11-04; First posted 2024-11-06 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Influenza Vaccines; Elderly
Keywords: influenza; adjuvanted vaccine; immunogenicity; elderly; safety
MeSH Terms: conditions — Influenza, Human | interventions — GBP510 vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- adjuvanted (Experimental): adjuvanted (aIIV4) influenza vaccine
  Interventions: Drug: adjuvanted
- non-adjuvanted (Active Comparator): non-adjuvanted (IIV4) influenza vaccine
  Interventions: Drug: non-adjuvanted

INTERVENTIONS:
Drug: adjuvanted — adjuvanted (aIIV4) influenza vaccine in the Taiwanses elderly with chronic medical conditions
  Arms: adjuvanted
Drug: non-adjuvanted — non-adjuvanted (IIV4) influenza vaccine in the Taiwanses elderly with chronic medical conditions
  Arms: non-adjuvanted

SUMMARY:
To compare the immunogenicity, cellular immune response, and safety between adjuvanted (aIIV4) and non-adjuvanted (IIV4) seasonal influenza vaccines in the Taiwanese elderly population with chronic medical conditions.

DETAILED DESCRIPTION:
Annual influenza vaccination is the most important and cost-effective intervention in reducing the impact of influenza, and a key component of the WHO response and preparedness efforts for influenza of pandemic potential. Reduced effectiveness of conventional egg-based vaccination was observed among risk group, such as elderly and people on with chronic medical conditions, which may result from their impaired immunogenicity. WHO, as well as ACIP of the USA, Europe, and Australia suggested adjuvanted influenza vaccines as one of alternatives for those people, which could decrease the disease burden significantly in several analyses. An adjuvanted commercial vaccine has been approved in Taiwan recently, but the local data of safety and effectiveness analysis is limited. This 1-year randomized control trial is designed to estimate the safety and effectiveness of adjuvanted influenza vaccine among Asian elderly people when compared to non-adjuvanted vaccines.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 65 years or above
* Presence of at least 1 chronic medical condition associated with increased risk of complicated influenza, including hypertension, chronic obstructive pulmonary disease (group A, B, E), asthma, congestive heart failure (ACC/AHA stage A, B, C, D), coronary arterial disease, diabetes mellitus, chronic liver disease (Child-Pugh score A, B, C) or chronic kidney disease (stage 1~4), neuromuscular disorders, hematological or solid organ malignancies, recipient of hematopoietic stem cell transplantation or solid organ transplantation.

Exclusion Criteria:

* Contraindications to influenza vaccination including history of severe adverse event after vaccination, such as anaphylaxis or Guillain-Barré Syndrome, or a severe bleeding tendency
* Prior receipt of influenza vaccination during the current flu season.
* Determination by the Principal Investigator (PI) that the participant is ineligible for enrollment based on clinical assessment.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-11-05 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The seroconversion rate (SCR) measured by the change in hemagglutination inhibition (HI) titer against the vaccine strains in serum between Day 1 (pre-vaccination) and Day 29. | Measured through Day 29
  The seroconversion rate (SCR) measured by the change in hemagglutination inhibition (HI) titer against the vaccine strains in serum between Day 1 (pre-vaccination) and Day 29.

SECONDARY OUTCOMES:
The geometric mean titer (GMT), seroprotection rate (SPR), cellular immune responses on Day1, Day 29 (±3), Day 181 (±7), and Day 361 (±7) | Measured through Day 361
  The geometric mean titer (GMT), seroprotection rate (SPR), cellular immune responses on Day1, Day 29 (±3), Day 181 (±7), and Day 361 (±7)
Incidence of severe adverse reactions within 28 days after immunization. | Measured through Day 28
  Incidence of severe adverse reactions within 28 days after immunization.
Incidence of laboratory-confirmed influenza during the study period. | Measured through Day 361
  Incidence of laboratory-confirmed influenza during the study period.
Incidence of emergency department visits and hospitalizations related to respiratory illness, all-cause mortality during the study period. | Measured through Day 361
  Incidence of emergency department visits and hospitalizations related to respiratory illness, all-cause mortality during the study period.

IPD SHARING:
Plan to Share IPD: Undecided